CLINICAL TRIAL: NCT05961267
Title: Study of Gynecological Follow-up of Patients With Autoimmune Disease or Inflammatory Rheumatism
Acronym: MARIGYN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/25
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Arthritis, Rheumatoid; Spondylitis, Ankylosing; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Sjogren's Syndrome; Mixed Connective Tissue Disease
Keywords: Auto-immune diseases; rare auto-immune diseases; contraception; gynecological follow-up
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Sjogren's Syndrome; Mixed Connective Tissue Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with a diagnosis of systemic lupus erythematosus, Gougerot-Sjögren's syndrome, scleroderma, Sharp's syndrome, rheumatoid arthritis or spondyloarthritis, according to current international standards.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — A gynecological follow-up questionnaire will be proposed to patients with one of the above mentioned pathologies. This is a standardized questionnaire specifically designed for this study.

SUMMARY:
Autoimmune diseases are the consequence of an abnormality of the immune system, leading it to attack components of our own body. They have a wide variety of presentations. They preferentially affect women, and often at a young age. Systemic lupus erythematosus, for example, most often occurs between the ages of 15 and 40.

Inflammatory rheumatism, such as spondyloarthritis or rheumatoid arthritis, is less prevalent in women, but also affects young people, and is particularly common.

Several disease-modifying treatments exist, depending on the severity and evolutivitý of the disease. Some are contraindicated or not recommended during pregnancy and therefore require supervision of pregnancy plans.

In addition, some treatments have an immunosuppressive activitý, which implies an annual screening of cervical lesions by cervico-uterine smear.

In this context, an adapted gynecological follow-up seems indispensable. The rheumatologist and the internist physician have a crucial role in advising and referring patients to their gynecological colleagues.

Studying the qualitý of this gynecological follow-up in a cohort of patients with autoimmune disease or inflammatory rheumatism is of major interest.

DETAILED DESCRIPTION:
To evaluate the gynecological follow-up of patients with autoimmune diseases or inflammatory rheumatism by:

* Assessing the proportion of patients reporting having contraception described as effective by guidelines within one year in the study population.
* Evaluating the proportion of patients reporting having had a consultation for screening or follow-up for cervical dysplasia in the year.

Descriptive analysis of :

* Factors associated with effective contraceptive use and frequency of cervical smear screening.
* The impact of the disease on the pregnancy project.
* The appropriateness of the chosen contraceptive and the patients' comorbidities.
* The prevalence of Human Papillomavirus (HPV) infections, cervical dysplasia, cervical cancer in this French population at risk.
* Barriers to gynecological care.

ELIGIBILITY:
Inclusion Criteria:

* Female patient over 18 years of age
* Non-menopausal patient (only for the subgroup of patients used to assess the use of effective contraception)
* Patient with a diagnosis of systemic lupus erythematosus, Gougerot-Sjögren's syndrome, scleroderma, Sharp's syndrome, rheumatoid arthritis or spondyloarthritis, according to current international standards.
* French-speaking patient with no comprehension problems
* Person affiliated with or benefiting from a social securitý scheme
* Patient who received information about the protocol and gavé her consent

Exclusion Criteria:

* Pregnant or breastfeeding patient
* Patient with a history of total hysterectomy
* Patient referred to in articles L 1121-5 to L 1121-8 (persons deprived of liberty by a judicial or administrative decision, minors, adults subject to a legal protection measure or unable to express their consent).

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patient with a diagnosis of systemic lupus erythematosus, Gougerot-Sjögren's syndrome, scleroderma, Sharp's syndrome, rheumatoid arthritis or spondyloarthritis, according to current international standards.
Sampling Method: Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who report having a screening of cervical dysplasia during the year according to international recommendations. | At baseline (Day 0)

SECONDARY OUTCOMES:
Proportion of patients who report using effective contraception during the year. | At baseline (Day 0)
Proportion of patients who report that their auto-immune pathology had an impact on their pregnancy plans. | At baseline (Day 0)
Proportion of patients whose contraception does not comply with recommendations regarding their comorbidities. | At baseline (Day 0)
Prevalence of HPV infections in the study sample. | At baseline (Day 0)
Prevalence of cervical dysplasia in the study sample. | At baseline (Day 0)
Prevalence of cervical cancer in the study sample. | At baseline (Day 0)
Proportion of patients who report not having consulted their gynecologist during the year. | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe RICHEZ, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de rhumatologie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No